CLINICAL TRIAL: NCT07286162
Title: Trauma-Focused Managing Cancer And Living Meaningfully (CALM-TF): A Phase III Randomized Controlled Trial of an Intervention Targeting Traumatic Stress in Patients With Advanced Ovarian Cancer
Brief Title: Trauma-Focused Managing Cancer And Living Meaningfully (CALM-TF) for Newly Diagnosed and Recurrent Ovarian Cancer
Acronym: CALM-TF
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Ovarian Cancer Canada (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OZUHN-045
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer (OvCa); Recurrent Ovarian Cancer
Keywords: randomized controlled trial; ovarian cancer; recurrence; newly diagnosed; CALM; Managing Cancer And Living Meaningfully; Psychotherapy; psychosocial support
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence

STUDY DESIGN:
Intervention Model Description: Participants randomized to the intervention arm of the trial will receive: Usual care, plus Trauma focused Managing Cancer and Living Meaningfully (referred to as CALM-TF), a psychotherapeutic intervention that aims to alleviate traumatic stress symptoms in patients with advanced cancer.
  Participants randomized to the control arm of the trial will receive: Usual care alone, which may include referral for psychosocial/psychiatric support should the patient request it, or should their clinician deem such support necessary. The trial team will not interfere with usual care referrals, but such referrals will be documented in the trial records.
Who Masked: Outcomes Assessor
Masking Description: Data analysts will also be blinded to participant treatment group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CALM-TF plus Usual Care (Experimental): Participants receive Trauma-Focused Managing Cancer and Living Meaningfully (CALM-TF), a brief manualized psychotherapeutic intervention consisting of 3-6 individual sessions over 3-6 months (45-60 minutes each). Sessions delivered via secure video conferencing (Microsoft Teams), telephone, or in-person based on participant preference. Participants also continue to receive usual standard of care throughout the intervention period.
  Interventions: Behavioral: Trauma-Focused Managing Cancer and Living Meaningfully
- Usual Care Alone (No Intervention): Participants receive usual standard of care only, which includes frequent conversations with their medical team regarding their care and meetings with social workers regarding financial or other practical issues. Participants have access to formal or specialized psychotherapeutic interventions upon referral by their primary physician or member of their circle of care.

INTERVENTIONS:
Behavioral: Trauma-Focused Managing Cancer and Living Meaningfully — CALM-TF is a brief, manualized psychotherapeutic intervention that incorporates trauma-focused elements into the established CALM framework. It includes a present-oriented focus with particular attention to affect regulation, relational support, and attachment security, specifically designed to address traumatic stress symptoms triggered by a diagnosis or recurrence.
  The intervention consists of 3-6 sessions delivered over 3-6 months, with each session lasting 45-60 minutes. Sessions are delivered by trained therapists through multiple modalities including secure web-conferencing software (Microsoft Teams), telephone, or in-person visits based on patient preference.
  CALM-TF focuses on four broad and interconnected content domains: (1) symptom management and communication with healthcare providers; (2) changes in self and in relationships with close others; (3) sense of meaning and purpose in life; and (4) hopes and fears about the future and mortal
  Other Names: CALM-TF
  Arms: CALM-TF plus Usual Care

SUMMARY:
The goal of this clinical trial is to investigate if CALM-TF (Trauma-Focused Managing Cancer and Living Meaningfully) is effective in treating traumatic stress symptoms in women with advanced ovarian cancer. It will also learn whether the efficacy differs at new diagnosis versus at recurrence.

The main questions it aims to answer are:

1. What is the effectiveness of CALM-TF in reducing traumatic stress symptoms in patients with newly diagnosed or recurrent advanced ovarian cancer, as measured at 3 and 6 months?
2. What are the effects of CALM-TF on depression, quality of life, and patient-perceived benefit of the intervention compared to usual care alone?
3. What are patient perceptions of their care experiences as explored through qualitative interviews?

Researchers will compare CALM-TF to usual standard of care (which includes regular conversations with medical teams and meetings with social workers) to see if CALM-TF works to treat traumatic stress.

Participants will:

* Receive 3-6 sessions of CALM-TF over 3-6 months (45-60 minutes each) via video call, telephone, or in-person based on preference, OR receive usual care only
* Complete questionnaires at baseline, 3 months, and 6 months
* Continue to receive their standard cancer care throughout the study
* Some participants may be invited to participate in qualitative interviews at 6 months

DETAILED DESCRIPTION:
This study examines whether a brief psychotherapy called Trauma-Focused Managing Cancer and Living Meaningfully (CALM-TF) can help women with advanced ovarian cancer who are experiencing traumatic stress symptoms.

Traumatic stress refers to the psychological impact of traumatic events, which in cancer care includes the diagnosis, progression, or recurrence of advanced disease. Research shows that up to 45% of patients with ovarian cancer experience clinically significant traumatic stress symptoms that meet diagnostic criteria for acute stress disorder.

CALM-TF is a manualized psychotherapeutic intervention that builds on an established therapy called CALM (Managing Cancer and Living Meaningfully), which has previously been shown to reduce depression and improve communication with healthcare providers in patients with advanced cancer. CALM-TF incorporates trauma-focused components specifically designed to address traumatic stress symptoms that arise at the time of diagnosis or recurrence of ovarian cancer.

The intervention consists of 3-6 individual therapy sessions delivered over 3-6 months, with each session lasting 45-60 minutes. Sessions can be conducted via secure video conferencing, telephone, or in-person based on participant preference. The therapy focuses on four interconnected content areas: symptom management and communication with healthcare providers; changes in self and relationships with close others; sense of meaning and purpose in life; and hopes and fears about the future and mortality, with trauma-focused components integrated throughout.

This is a multi-site randomized controlled trial enrolling 300 women with newly diagnosed stage III or IV ovarian cancer or recurrent ovarian cancer (within six months of diagnosis or recurrence). Participants are randomly assigned in a 1:1 ratio to receive either CALM-TF plus usual care or usual care alone. Usual care includes regular conversations with medical teams and meetings with social workers regarding financial or practical issues, with access to specialized psychological support through referral.

The study uses validated questionnaires to measure traumatic stress symptoms, depression, quality of life, death anxiety, and perceived benefit of care at three time points: baseline, 3 months, and 6 months after enrolment. The primary outcome is traumatic stress symptoms at 6 months measured by the Stanford Acute Stress Reaction Questionnaire-II (SASRQ-II), a 30-item instrument with scores ranging from 0-150, where scores above 40 indicate clinically significant symptoms.

A subset of up to 30 participants will be invited to participate in qualitative interviews after completing their 6-month assessment to share their experiences with the intervention or usual care, explore factors that influenced their traumatic stress experience, and discuss how the therapy was integrated into their daily lives. The study also includes a health economic evaluation to assess the cost-effectiveness of CALM-TF compared to usual care over the 6-month period.

The findings of this RCT will inform healthcare policy and clinical practice guidelines for comprehensive psychosocial care, with potential for CALM-TF to be integrated into standard care.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed stage III or IV ovarian cancer OR recurrent ovarian cancer within six months of diagnosis or recurrence
* Age 18 years or older
* Able to speak and read English
* Able to provide informed consent

Exclusion Criteria:

* Significant cognitive impairment that would interfere with the ability to participate in psychotherapy or complete study questionnaires
* Active psychosis or severe psychiatric condition requiring immediate psychiatric intervention
* Receiving ongoing psychotherapy at the time of recruitment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2031-03-01 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Stanford Acute Stress Reaction Questionnaire-II (SASRQ-II) | From enrolment to the end of study at 6 months
  Traumatic stress symptoms are measured by the Stanford Acute Stress Reaction Questionnaire-II (SASRQ-II), a validated 30-item self-report instrument specifically designed to assess traumatic stress symptoms based on DSM-5 criteria. The SASRQ-II provides a total score range of 0-150, where higher scores reflect increasing symptom severity and cut-off scores of >40 indicate clinically significant traumatic stress symptoms.

SECONDARY OUTCOMES:
Experiences in Close Relationships-Modified-16 (ECR-M-16) | Baseline only
  Attachment security is measured by the ECR-M-16, a validated 16-item measure adapted to measure close relationships in patients with advanced cancer. Two 8-item subscales are derived from this measure, reflecting levels of anxious attachment and avoidant attachment, which can be helpful to understand and address attachment issues in patients with advanced cancer. Items are rated from 1 (agree) to 7 (disagree), with higher scores reflecting greater attachment insecurity.
Condensed Memorial Symptom Assessment Scale (CMSAS) | From enrolment to the end of the study at 6 months
  Physical symptoms commonly experienced by cancer patients are measured by the Condensed Memorial Symptom Assessment Scale (CMSAS), a validated 14-item instrument that assesses distress related to symptoms including pain, fatigue, nausea, and drowsiness. Serves as an important covariate to control for physical symptom burden that may influence psychological outcomes. Symptoms are rated as present or not, with the level of distress associated with physical symptoms rated from 0 (not at all) to 4 (very much), and the frequency of psychological symptoms (worry, feeling sad, feeling nervous) rated 1 (rarely) to 4 (almost constantly). Higher scores reflect increasing symptom burden.
Patient Health Questionnaire (PHQ-9) | From enrolment to the end of the study at 6 months
  Depression severity is measured by the Patient Health Questionnaire (PHQ-9), a validated 9-item instrument assessing depression severity that has demonstrated reliability and validity in cancer populations. Scores may range from 0-27, with higher scores reflecting increasing severity of depressive symptoms. A cut-off score of 10 is used to reflect moderate depressive symptoms.
Death and Dying Distress Scale (DADDS) | From enrolment to the end of the study at 6 months
  Distress related to thoughts on death and dying are measured by the Death and Dying Distress Scale (DADDS), a validated 15-item questionnaire evaluating distress caused by a patient's thoughts on death and dying. Factor analysis demonstrates distress related to two factors: Finitude and Dying. Total scores may range from 0-75, with higher scores indicating greater death-related distress.
EuroQol 5-Dimension 5-Level Health Questionnaire (EQ-5D-5L Health Questionnaire) | From enrolment to the end of the study at 6 months
  Health-related quality of life is measured by the EQ-5D-5L Health Questionnaire, a validated instrument that measures quality of life across five dimensions (mobility, self-care, activities, pain, and anxiety) using a 5-level scale. It provides both a health state profile and a single utility index value. Dimension scores are rated from 1 (no problems) to 5 (extreme problems), with higher scores reflecting worse health status. The single utility index score is rated from 0 (worst imaginable health) to 100 (best imaginable health).
Short Form 6-Dimensions Health Survey (SF-6D Health Survey) | From enrolment to the end of the study at 6 months
  Health-related quality of life is measured by the SF-6D Health Survey, derived from the Short Form-36 health questionnaire. It evaluates six health dimensions (physical functioning, role limitations, social functioning, pain, mental health, and vitality), each rated from 0 (worst health state, e.g. death) to 1.0 (best health state, e.g., full health). This measure also allows for the calculation of quality adjusted life years (QALYs), which can be used to evaluate cost-effectiveness of health care interventions.
Clinical Evaluation Questionnaire (CEQ) | At 3 and 6 month time points.
  Perceived benefit of interactions with healthcare providers are measured by the Clinical Evaluation Questionnaire (CEQ), a validated 7-item patient-reported experience questionnaire that assesses perceived benefit in domains relevant to advanced cancer, including patient-provider communication and perceived quality of care. Items are rated on perceived helpfulness of the interactions, ranging from 0 (not at all) to 4 (very much), with an option to answer 'not applicable'. A total score is calculated by summing the item scores; 'not applicable' responses are considered missing data. Higher scores reflect greater perceived benefit of the interactions with healthcare providers.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lheureux, MD, PhD, Principal Investigator — Princess Margaret Cancer Centre, University Health Network; Gary Rodin, MD, Principal Investigator — Princess Margaret Cancer Centre, University Health Network
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
The data sharing plan for this study has not yet been finalized. Decisions regarding individual participant data (IPD) sharing will be made in consultation with the study sponsor, institutional policies, and applicable regulations. Any data sharing would occur only after completion of primary analyses and would require appropriate data use agreements to protect participant privacy and confidentiality. The study team will consider requests for de-identified data from qualified researchers for purposes of meta-analyses or secondary research questions aligned with the original study aims.